CLINICAL TRIAL: NCT05424471
Title: Preventing Early Childhood Obesity, Part 1: Family Spirit Nurture, 3-9 Months, Long-term Follow-up
Brief Title: Preventing Early Childhood Obesity, Part 1: Long-term Follow-up
Acronym: PECO1-LTF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 7476 /MOD994
Record Dates: First submitted 2022-04-26; First posted 2022-06-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Obesity; Water; Lack of; Childhood Obesity; Feeding Behavior; Mother-Child Relations; Dietary Habits
Keywords: Sugar Sweetened Beverages
MeSH Terms: conditions — Obesity; Pediatric Obesity; Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Family Spirit Nurture (FSN) (Experimental): Intervention group participants receive 1 Family Spirit Nurture lesson taught by Family Health Coaches. Mothers will receive the lesson within 1-2 weeks of completing the 4-year Follow-up Assessment. The lesson focuses on age-appropriate parental feeding practices, including snack routines, avoidance of SSBs and promotion of water consumption. The lesson is highly visual and interactive, and incorporates cultural teachings related to child feeding and nutrition that support aims. The Family Health Coaches also provide social support and will facilitate referrals to community resources.
  Interventions: Behavioral: Family Spirit Nurture (FSN)
- Control Vehicle Safety (Other): Control group participants receive 1 lesson with vehicle safety information, taught by Family Health Coaches. Mothers will receive the lesson within 1-2 weeks of completing the 4-year Follow-up Assessment. The Family Health Coaches also provide social support and will facilitate referrals to community resources.
  Interventions: Other: Control Group - Vehicle Safety

INTERVENTIONS:
Behavioral: Family Spirit Nurture (FSN) — The FSN intervention lesson is taught to participants previously randomized into the FSN intervention group during the PECO 1 study. Intervention group participants receive 1 Family Spirit Nurture lesson taught by Family Health Coaches. Mothers will receive the 1 - 45 minute lesson within 1-2 weeks of completing the 4-year Follow-up Assessment. The lesson focuses on age-appropriate parental feeding practices, including snack routines, avoidance of SSBs and promotion of water consumption. The lesson is highly visual and interactive, and incorporates cultural teachings related to child feeding and nutrition that support aims. The Family Health Coaches also provide social support and will facilitate referrals to community resources.
  Arms: Family Spirit Nurture (FSN)
Other: Control Group - Vehicle Safety — The control (vehicle safety) lesson is taught to participants previously randomized into the control group during the PECO 1 study. Control group participants receive 1 - 30 minute lesson with vehicle safety information, taught by Family Health Coaches. Mothers will receive the lesson within 1-2 weeks of completing the 4-year Follow-up Assessment. The Family Health Coaches also provide social support and will facilitate referrals to community resources.
  Other Names: Vehicle Safety
  Arms: Control Vehicle Safety

SUMMARY:
This study extends follow up on of Native American (NA) mothers and their children (now age 3-5 years) enrolled in the 1:1 randomized controlled trial of the Family Spirit Nurture (FSN) intervention designed to prevent early childhood obesity (PECO 1). The investigators will examine whether positive FSN impacts on sugar sweetened beverage (SSB) consumption and healthy growth in the first year of life were sustained. The investigators will also examine the effects of the emergency COVID-19 water solutions on water insecurity, early childhood SSB consumption, and growth, and explore how COVID-19 affected child feeding patterns and weight status either through changes in maternal mental health or household food access.

DETAILED DESCRIPTION:
Primary Aims

Aim 1. Determine the longer-term effectiveness of the brief FSN intervention on reducing SSB consumption, increasing water intake, and promoting healthy growth status up to 5 years of age.

Aim 2. Examine the impact of point-of-use (POU) water filters, employed as COVID-19 emergency water response efforts, on water insecurity, children's water intake and SSB consumption with or without previous FSN intervention. Positive findings would provide leverage to promote water solutions and water equity.

Secondary Aims

Secondary Aim 1. Determine whether providing a booster lesson at 4 years of age targeting age appropriate parental feeding practices, snack routines, avoidance of SSBs and increased water intake impacts SSB consumption and water intake between 4 and 4.5 years of age and child growth between 4 and 5 years of age.

Secondary Aim 2. Describe how COVID-19 affected child feeding patterns and weight status either through maternal depression and anxiety or changes in food access.

This follow-up study will builds upon a 1:1 randomized controlled trial of the Family Spirit Nurture (FSN) intervention designed to prevent early childhood obesity (PECO 1).

Methods:

A long-term follow-up evaluation will be conducted with n=110 of the randomized mother-child dyads (90% of the participants that completed the PECO 1 study) when the children are between 4 - 5 years of age.

Eligible participants will complete a 4 year follow-up assessment after reconsent when the children are 4 years of age. All participants will maintain their randomization status and receive one age appropriate lesson specific to their study group. The intervention group (n=55) will receive one FSN lesson focused on age-appropriate parental feeding practices, including snack routines, avoidance of SSBs, and increased water intake. The control group (n=55) will receive one injury prevention lesson focused on vehicle safety. An endline follow-up assessment will be completed by all reconsented participants after three months of the 4 year follow-up assessment. Maternal and child medical chart review will be conducted by trained study staff after the child turns 5 years old. Medical chart reviews will collect data on maternal BMI (as a possible moderator of child growth) and child growth.

During the COVID-19 pandemic as part of the emergency response on the Navajo Nation, a subset of study participants who previously reported water insecurity (n=50) received point-of-use (POU) water filters. Water filters were evenly distributed between the intervention (n=25) and control groups (n=25).

Study implementation will include three phases:

Phase 1 (Reconsent, Reenroll, and 4 year Follow-up Assessment):

Study staff will re-approach randomized mother/child dyads when the child is 4 years of age to complete the informed consent process for the follow-up component. Participants will maintain their original randomization status and complete a 4 year follow-up assessment that consists of a mixed-methods approach.

Phase 2 (Booster Lesson):

Local FHCs, trained and employed by Johns Hopkins, will deliver either the intervention (1- FSN lesson) or the control condition (1- Vehicle-Safety Lesson) shortly after the 4 year follow-up assessment when the child is 4 years of age. With participant permission, lesson visits will be audio recorded for quality assurance, using digital audio recorders. A random 10% of audio recordings will be reviewed and rated to ensure fidelity to the curriculum and to facilitate staff training and supervision.

Phase 3 (Endline Follow-up Assessment and Medical Chart Reviews):

Three months after the 4 year follow-up assessment, participants will complete an endline follow-up assessment. The endline follow-up assessment will be the same assessment battery as the 4 year follow-up assessment. Maternal and child medical chart reviews will be conducted by trained study staff after the child is 5 years of age. Weight and height data will be collected from child's medical charts (birth through 5 years of age). Data may be collected any time during the 5th year of life as timing of the five year check up can vary. Maternal BMI will be collected from maternal medical chart reviews as a possible moderator of child growth.

ELIGIBILITY:
Inclusion Criteria:

* Mother/child dyads who enrolled, participated in/completed the initial PECO 1 study (followed mother/infant dyads through 12 months of age).
* Willingness to fully participate.

Exclusion Criteria:

* Inability to participate in full intervention or evaluation (e.g., planned move, etc.)

Min Age: 13 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 110 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Group differences in children's mean BMI z-scores over time as assessed through child weight and length/height measurements through 5 years of age. | Birth to 5 years of age
  Child weight (to the nearest ounce) and recumbent length/height (to the nearest 1/8 inch) will be extracted through medical chart review. Measurements will be taken by healthcare providers. Measurements will be used to calculate BMI z-scores using age- and sex-specific World Health Organization (WHO) Child Growth Standards.
Group differences in sugar sweetened beverage (SSB) consumption & water intake. | 3 months to 5 years of age
  Mothers were asked about SSB initiation and frequency among infants between 3 months and 12 months of age in the Preventing Early Childhood Obesity, Part 1: Family Spirit Nurture, 3-9 Months study using an an adapted version of the Pre-School-Aged Beverage Intake Questionnaire (BEVQ-15). We will continue to use the age appropriate Pre-School-Aged BEVQ-15 to assess child's SSB consumption and water intake between 4 and 5 years of age. This data will be examined for between group differences in SSB consumption and water intake through 5 years of age.
Examine whether point-of-use (POU) water filters impact water security, and/or moderate intervention impact on water intake and SSB consumption. | 3 to 5 years of age
  Examine the impact of point-of-use (POU) water filters, employed as COVID-19 emergency water response efforts, on water insecurity. Examine study group differences in water intake and SSB consumption with and without POU water filters.

SECONDARY OUTCOMES:
Between study group differences, post booster lesson, in age appropriate parental feeding practices, snack routines, avoidance of SSBs and increased water intake. | Up to 5 years of age
  Age appropriate parental feeding practices, snack routines, avoidance of SSBs and increased water intake impacts SSB consumption and water intake between 4 and 4.5 years of age will be measured by the Toddler BEV-Q and Child Feeding Styles Questionnaire. Child growth between 4 and 5 years of age will be assessed by weight and length/height measurements from medical chart reviews.
Within study group comparison of pre-/during- COVID-19 child feeding practices, snack routines, SSB consumption and water intake and examination of associations with maternal depression and anxiety, and changes in food access. | 5 years postpartum
  COVID-19 Impact Questionnaire will be used to assess how the COVID-19 pandemic has affected participants' lives, access to basic needs and healthcare, child feeding practices and childcare support. The Toddler BEV-Q and Child Feeding Styles Questionnaire will be used to assess child feeding practices, snack routines, SSB consumption and water intake. Maternal depression will be assessed by the CES-D and anxiety will be assessed by PROMIS Anxiety 8-item scale.

CONTACTS AND LOCATIONS:
Overall Officials: Allison Barlow, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins Center for American Indian Health, Shiprock, New Mexico, United States